CLINICAL TRIAL: NCT03527082
Title: Women's Knowledge and Attitudes to Use of Mesh in Gynaecological Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Epsom and St Helier University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 241922
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-01

CONDITIONS: Prolapse, Vaginal
Keywords: mesh; erosion; transvaginal; prolapse; laparoscopic; tension free tape
MeSH Terms: conditions — Uterine Prolapse; Prolapse | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women attending gynaecology clinics: 150 women attending gynaecology clinics that fulfil inclusion criteria
  Inclusion criteria:
  Inclusion criteria
  1. Over the age of 18
  2. attending gynaecology clinics
  3. Able to read and comprehend the details of the study in patient information sheet.
  4. Mentally competent at signing the consent form.
  5. English -speaking, if not then translator available
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire of 20 items evaluating attitudes and perception of mesh use in gynaecological surgery. Questionnaire will take 10 minutes to complete. For non-English speaking patients a translator will be sought, where feasible to help women complete the questionnaire.
  Participation will be entirely voluntary and also the questionnaire will be piloted to ensure that questions asked are clear and concise. Questionnaire is anonymised and does not contain patient identifying information thereby eliminating breach of confidentiality.

SUMMARY:
This is a questionnaire study that is being performed to ascertain the knowledge and attitudes of women towards use of mesh in gynaecological surgery. Women over the age of 18, able to read and comprehend the information leaflet, sign and give informed consent will be eligible to participate. Women who are not fluent in English will be able to participate if a translator can convey the information. The trial will be conducted at Epsom and St Helier Hospitals, in the United Kingdom. The investigators aim to recruit 150 women to this study. No power calculation has been performed as this is an exploratory study.

However, previous studies have included 64 and 77 women respectively.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) and stress urinary incontinence (SUI) are common conditions experienced by women. It is estimated that 20% of women undergo surgery for the treatment of prolapse. Transvaginal placement of surgical mesh for repair of POP and SUI are associated with complications such as erosion, infection, dyspareunia, bowel and bladder perforation as well as failure of the operation. Such complications have resulted in the FDA reclassifying transvaginal meshes to high risk medical devices. Most recently, National Institute for Clinical Excellence (NICE) in the United Kingdom has limited the use of transvaginal meshes for anterior and posterior compartment prolapse to a research context only.

Since the FDA and NICE publications, there has been much controversy and increasing litigation arising from complications of transvaginal mesh use. Recent negative media attention has likely affected patients' perception regarding mesh use in gynaecology. There are no studies assessing the knowledge and perception of mesh use in gynaecological surgery within the United Kingdom. Previous studies have found patients have limited knowledge and often are misinformed. However, these have been limited to transvaginal meshes. Laparoscopic procedures using mesh for POP such as sacrohysteropexy and sacrocolpopexy are become increasingly popular with comparable outcomes to vaginal surgery. The risk of mesh erosion with laparoscopic surgery is less than vaginal placement.

The use of mesh of gynaecology remains a topical issues and given the amount of information available to patients, this concept merits study, as it may influence patients' decision making and therefore a prominent part of the consent process. The use of mesh in gynaecological surgery remains a highly effective method of treating POP and SUI in appropriately selected patients and routes. It is therefore important to understand patients' understanding and perception regarding mesh use and sources of information in the wake of media coverage and attention. The investigators seek to evaluate patients' knowledge and attitudes towards use of mesh in gynaecological surgery presenting to gynaecology clinics.

The investigators aim to survey 150 women attending gynaecology clinics using a questionnaire. A power calculation has not been performed however, similar studies have included 164 and 77 women respectively. The questionnaire consists of 20 questions that should take 10 minutes to complete.

Consent: A valid consent with detailed written information sheet will be sought before including them in this trial.

Inclusion and exclusion criteria: All women attending the clinic will be eligible to participate if they are over the age of 18, with an understanding of English or translator available and able to provide informed consent.

Risks and benefits: All women will receive the same standard of care regardless if they agree to disagree to participate in the trial. There are no disadvantages associated with participation in taking part in the study.

Data storage: All the information obtained from this study will be stored in a confidential manner and will only be available to the researchers for future analysis.Participants can withdraw their consent at any point and this will not affect the standard of care given to them in future.All the information pertaining to the trial will be destroyed securely.

This research does not involve any use, storage of any tissue

ELIGIBILITY:
Inclusion Criteria:

* a. Women > 18 years of age attending gynaecology clinics

  b. Able to read and comprehend the details of the study in patient information sheet.

  c. Mentally competent at signing the consent form.

Exclusion Criteria:

1. Patient refusal.
2. Inability to consent due to a language barrier (no translator available, medication)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients attending gynaecology clinic
Study Population: Women attending gynaecology outpatient clinics at Epsom and St Helier's University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Women's Knowledge and Attitudes to Use of Mesh in Gynaecological Surgery | Duration of study, 12 months
  Assessed by use of questionnaire

REFERENCES:
- [Background] Brown LK, Fenner DE, Berger MB, Delancey JO, Morgan DM, Patel DA, Schimpf MO. Defining patients' knowledge and perceptions of vaginal mesh surgery. Female Pelvic Med Reconstr Surg. 2013 Sep-Oct;19(5):282-7. doi: 10.1097/SPV.0b013e31829ff765. PMID 23982577
- [Background] Dallenbach P, De Oliveira SS, Marras S, Boulvain M. Incidence and risk factors for mesh erosion after laparoscopic repair of pelvic organ prolapse by lateral suspension with mesh. Int Urogynecol J. 2016 Sep;27(9):1347-55. doi: 10.1007/s00192-016-2974-z. Epub 2016 Feb 17. PMID 26886554
- [Background] Dessie SG, Hacker MR, Haviland MJ, Rosenblatt PL. Attitudes toward transvaginal mesh among patients in a urogynecology practice. Int Urogynecol J. 2015 Jun;26(6):865-73. doi: 10.1007/s00192-014-2607-3. Epub 2015 Jan 17. PMID 25595568
- [Background] Iglesia CB. Synthetic vaginal mesh for pelvic organ prolapse. Curr Opin Obstet Gynecol. 2011 Oct;23(5):362-5. doi: 10.1097/GCO.0b013e32834a92ab. PMID 21857223
- [Background] Maher C, Feiner B, Baessler K, Schmid C. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD004014. doi: 10.1002/14651858.CD004014.pub5. PMID 23633316
- See also: National Institute for Health and Care Excellence. Transvaginal meshes for anterior and posterior prolapse. 2017 — http://www.nice.org.uk/guidance/ipg599/chapter/1-Recommendations